CLINICAL TRIAL: NCT03981640
Title: Neurovascular Control of Renal Blood Flow During Exercise in African American Adults
Brief Title: Neural Control of Kidney Blood Flow During Exercise in African American Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rachel Drew, Associate Professor, University of Massachusetts, Boston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1614; 1R15HL152359-01A1 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Exercise; Cold stress; Mental stress
MeSH Terms: conditions — Motor Activity; Stress, Psychological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African American Adults (Experimental): African American adults will undergo the interventions of acute exercise, a cold pressor test, and a mental stress test while beat-to-beat renal blood flow velocity, mean arterial blood pressure, and heart rate are recorded.
  Interventions: Other: Acute exercise; Other: Cold pressor test; Other: Mental stress test
- White Adults (Experimental): White adults will undergo the interventions of acute exercise, a cold pressor test, and a mental stress test while beat-to-beat renal blood flow velocity, mean arterial blood pressure, and heart rate are recorded.
  Interventions: Other: Acute exercise; Other: Cold pressor test; Other: Mental stress test

INTERVENTIONS:
Other: Acute exercise — Participants will lie in a semi-supine position with their feet attached to the pedals of a custom-arranged cycle ergometer. Participants' 40% heart rate reserve will be calculated, giving the target value to achieve during exercise based on appropriate resistance applied on the cycle ergometer, corresponding to a moderate exercise intensity. After a 5-minute resting baseline, participants will perform dynamic cycling exercise at steady state for up to 20 minutes. They will then stop exercising, and there will be a 5-minute recovery period. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. A rating of perceived exertion will be taken from participants during the last 30 seconds of steady-state cycling exercise.
Other: Cold pressor test — Participants will lie in a semi-supine position, and after a 3-minute resting baseline, participants will have their hand immersed in ice water for 2 minutes. This cold pressor test represents the non-exercise, physical sympathetic stressor. Participants' hand will then be removed from the ice water, followed by a 3-minute recovery period. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. Ratings of hand pain and cold perception will be taken from participants during the last 30 seconds of the cold pressor test.
Other: Mental stress test — Participants will lie in a semi-supine position, and after a 3-minute resting baseline, participants will perform a mental arithmetic task for 5 minutes. This mental stress test represents the non-exercise, psychological sympathetic stressor. Participants will be instructed to subtract a given number from a randomly selected three-digit number and verbally state their answer and continue to do so for the duration of the test. Participants will be instructed to state their answers as quickly and accurately as possible. Participants will then stop the arithmetic task, and a 3-minute recovery period will follow. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. A rating of perceived stress will be taken from participants during the last 30 seconds of the mental stress test.

SUMMARY:
The goal of this clinical trials is to learn if healthy young African American (AA) adults have a larger change in their kidney blood flow during exercise compared to White (W) adults. The main questions that this study aims to answer are:

* Do healthy young AA adults have a larger decrease in kidney blood flow during exercise compared to W adults?
* Do healthy young AA adults have a larger decrease in kidney blood flow during other types of stress compared to W adults?

During two visits in the research lab, participants will:

* Perform a fitness test
* Perform cycling exercise while lying down
* Undergo a cold hand test
* Perform a mental math test

Completing this clinical trial will help researchers to understand more about why many AA adults have heart and kidney problems, so future research can study ways to reduce the number of AA adults who have these health issues.

DETAILED DESCRIPTION:
African American (AA) adults have a greater prevalence of developing cardiovascular and renal disease (CVRD) than White (W) adults. Elevated sympathetic nervous system activity is associated with increased incidence of CVRD. Physical exertion, such as exercise, acutely increases sympathetic nervous system activity directed towards the kidneys, resulting in renal vasoconstriction and reduced renal blood flow (RBF). Limited research shows that healthy young AA adults exhibit exaggerated sympathetic responsiveness both at rest and during sympathetic activation, which may be a major contributor to the increased risk of CVRD in this population. However, the acute renal vasoconstrictor response to any sympathetic nervous system activation has not been investigated to date in AA adults. During sympathetic nervous system activation such as exercise, sympathetic outflow to the kidneys in AA adults might be exaggerated, contributing to greater renal vasoconstriction and a larger reduction in RBF. Over time, this exaggerated neurovascular response to sympathetic activation could have a negative cumulative effect on the kidneys, which could be a contributing factor to the greater incidence of CVRD in this population.

Therefore, this study aims to examine the renal vasoconstrictor response to sympathetic stressors in healthy AA adults prior to development of CVRD, which will be achieved via two Specific Aims. In Specific Aim 1, the investigators will test the hypothesis that the renal vasoconstrictor response to acute dynamic exercise is exaggerated in healthy young AA compared to W adults. Specifically, the investigators will measure RBF and blood pressure at rest and during cycling exercise to calculate renal vascular resistance responses to exercise, enabling us to test the hypothesis that healthy young AA adults exhibit an exaggerated renal vasoconstrictor response to acute cycling exercise compared to healthy young W adults. In Specific Aim 2, the investigators will test the hypothesis that the renal vasoconstrictor response to non-exercise sympathetic stressors is exaggerated in healthy young AA compared to W adults. Specifically, the investigators will measure RBF and blood pressure at rest and during a cold pressor and mental stress tests to calculate renal vascular resistance responses to these non-exercise sympathetic stressors, enabling us to test the hypothesis that healthy young AA adults exhibit exaggerated renal vasoconstrictor responses to non-exercise sympathetic stressors compared to healthy young W adults.

Using the highly innovative approach of Doppler ultrasound to measure RBF during exercise and non-exercise sympathetic stressors non-invasively and with high temporal resolution will enable us to assess the renal vasoconstrictor response to sympathetic stressors in healthy AA adults prior to development of CVRD, so the underlying integrative physiological responses to sympathetic activation in AA adults can be understood. Findings from this study in this understudied yet clinically significant area will contribute to the ultimate goal of creating and implementing treatment strategies to reduce the risk of developing CVRD in AA adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-report as either African American or White racial identity
* Born in United States
* Both biological parents identify as same racial identity as participant
* Recreationally active (participating in physical activity for at least 20 minutes per day, at least three times per week, but not training for competitive events)
* Fluent in English

Exclusion Criteria:

* Hispanic or Latino
* Females who are pregnant or lactating
* Cardiovascular or renal disease
* Hypertension (blood pressure of more than or equal to 130/80 mmHg)
* Diabetes
* Obesity (body mass index of more than or equal to 30 kg/m2)
* Smoker/Tobacco user
* Acute medical conditions
* Taking prescribed cardiovascular, antihypertensive, or renal medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male and female
Enrollment: 32 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in renal vascular resistance during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the percent change from pre-acute exercise to during steady-state exercise will be assessed.
Change in renal vascular resistance during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the percent change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in renal vascular resistance during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the percent change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.

SECONDARY OUTCOMES:
Change in renal blood flow velocity during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in mean arterial blood pressure during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in systolic blood pressure during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in diastolic blood pressure during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in heart rate during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in cardiac output during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in stroke volume during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in total peripheral resistance during acute exercise | Pre-acute exercise and during steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in renal blood flow velocity during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in mean arterial blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in systolic blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in diastolic blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in heart rate during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in cardiac output during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in stroke volume during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in total peripheral resistance during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in renal blood flow velocity during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in mean arterial blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in systolic blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in diastolic blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in heart rate during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in cardiac output during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in stroke volume during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in total peripheral resistance during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.

OTHER OUTCOMES:
Rating of perceived exertion during acute exercise | During last 30 seconds of steady-state exercise
  For the acute exercise intervention, the rating will be taken during the last 30 seconds of steady-state exercise. The Borg Scale of Perceived Exertion will be used, with which a rating from 6 to 20 will be taken, with 6 representing no exertion and 20 representing maximal exertion.
Rating of hand pain during cold pressor test | During last 30 seconds of cold pressor test
  For the cold pressor test intervention, the rating will be taken during the last 30 seconds of the cold pressor test. A scale from 0 to 10 will be used to take the rating, with 0 representing no pain and 10 representing the worst possible pain.
Rating of cold perception during cold pressor test | During last 30 seconds of cold pressor test
  For the cold pressor test intervention, the rating will be taken during the last 30 seconds of the cold pressor test. A scale from 0 to -11 will be used to take the rating, with 0 representing no perceived cold and -11 representing unbearable cold.
Rating of perceived stress during mental stress test | During last 30 seconds of mental stress test
  For the mental stress test intervention, the rating will be taken during the last 30 seconds of the mental stress test. A scale from 0 to 4 will be used to take the rating, with 0 representing no perceived stress and 4 representing extremely stressful.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C Drew, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No